CLINICAL TRIAL: NCT01388218
Title: Non-interventional Cross-over Study to Reduce Items of the Draft PROactive Tools as a Measure of Physical Activity in Daily Life in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Non-interventional Cross-over Study to Reduce Items of PROactive Tools Measuring Physical Activity in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: KU Leuven (Other); University of Edinburgh (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); University Medical Center Groningen (Other); University of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: PROactive WP4
Record Dates: First submitted 2011-07-04; First posted 2011-07-06 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Physical Activity; Patient Reported Outcome (PRO); Chronic obstructive pulmonary disease (COPD); Innovative Medicines Initiative - Joint Undertaking (IMI-JU)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Arm 1 - Daily+Clinical: Order of assessment: Daily PRO + Clinical visit PRO
- Arm 2 - Clinical+Daily: Order of assessment: Clinical visit PRO + Daily PRO

SUMMARY:
The purpose of the protocol is to develop final draft PRO instruments of physical activity in daily life to be used and evaluated in the further validation studies measuring physical activity in chronic obstructive pulmonary disease (COPD) patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria: post bronchodilator forced expiratory volume in one second (FEV1)/forced vital capacity (FVC)<70%) confirmed with spirometry in stable clinical conditions. For patients recruited during an exacerbation, the diagnosis of COPD should be confirmed in stable conditions.
* Current or ex-smokers with a smoking history equivalent to at least 10 pack years.
* Able to read and write and to use electronic devices and physical activity monitor.

Exclusion Criteria:

* Orthopaedic, neurological or other complaints that significantly impair normal biomechanical movement patterns, as judged by the investigator.
* Respiratory diseases other than COPD (e.g. asthma).
* Cognitive impairment, as judged by the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable COPD patients from Outpatients clinics and Primary care clinic
  Exacerbated COPD patients from Inpatients
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Garcia-Aymerich, MD, PhD, Study Chair — Barcelona Institute for Global Health; Niklas Karlsson, Study Chair — AstraZeneca; Thierry Troosters, Principal Investigator — KUL Leuven; Thys van der Molen, Principal Investigator — University Medical Center Groningen; Nick Hopkinson, MD, Principal Investigator — Imperial College London; Roberto Rabinovich, MD, PhD, Principal Investigator — University of Edinburgh; Ioannis Vogiatzis, PhD, Principal Investigator — Thorax Research Foundation Athens
Locations (5):
- University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Leuven, Belgium
- Thorax Research Foundation, Athens, Greece
- University Medical Center, Groningen, Netherlands
- United Kingdom (2):
  - Royal Brompton Hospital, Imperial College, London, England
  - ELEGI/Colt laboratory UoE/MRC Centre for Inflammation Research The Queen's Medical Research Institute, University of Edinburgh, Edinburgh, Scotland

REFERENCES:
- [Result] Gimeno-Santos E, Raste Y, Demeyer H, Louvaris Z, de Jong C, Rabinovich RA, Hopkinson NS, Polkey MI, Vogiatzis I, Tabberer M, Dobbels F, Ivanoff N, de Boer WI, van der Molen T, Kulich K, Serra I, Basagana X, Troosters T, Puhan MA, Karlsson N, Garcia-Aymerich J; PROactive consortium. The PROactive instruments to measure physical activity in patients with chronic obstructive pulmonary disease. Eur Respir J. 2015 Oct;46(4):988-1000. doi: 10.1183/09031936.00183014. Epub 2015 May 28. PMID 26022965
- [Derived] Demeyer H, Gimeno-Santos E, Rabinovich RA, Hornikx M, Louvaris Z, de Boer WI, Karlsson N, de Jong C, Van der Molen T, Vogiatzis I, Janssens W, Garcia-Aymerich J, Troosters T, Polkey MI; PROactive consortium. Physical Activity Characteristics across GOLD Quadrants Depend on the Questionnaire Used. PLoS One. 2016 Mar 14;11(3):e0151255. doi: 10.1371/journal.pone.0151255. eCollection 2016. PMID 26974332
- See also: Related Info — http://www.proactivecopd.com